CLINICAL TRIAL: NCT01127984
Title: Pocket Haematoma Prevention in Patients Who Required Implantation/Replacement of a Pacemaker or Implantable Cardiac Defibrillator (ICD) During Dual Antiplatelet or Anticoagulant Therapy. A Prospective Randomized Trial. The PHP Study.
Brief Title: Pocket Haematoma Prevention in Patients Who Required Implantation/Replacement of a Pacemaker or Implantable Cardiac Defibrillator. The PHP Study.
Acronym: PHP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Careggi Hospital (Other)
Responsible Party: Emilio Vincenzo Dovellini, MD, Careggi Hospital, Division of Invasive Cardiology 1, Florence, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOVE 1
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2010-05

CONDITIONS: Pacemaker Implantation; Pocket Hematoma and Bleeding; Antiplatelet Therapy or Oral Anticoagulants
Keywords: pacemaker; pocket haematoma; antiplatelet therapy; fibrin glue
MeSH Terms: conditions — Hemorrhage | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment with tissucol (Experimental): patients treated with tissucol, local application in the pocket of PM / ICD
  Interventions: Drug: tissucol
- vacuum drainage system (Active Comparator): patients treated with application of vacuum drainage system.
  Interventions: Procedure: drainage system

INTERVENTIONS:
Drug: tissucol — dosage: 2 or 5 ml Frequency: 1 application Duration: 5 minutes
  Other Names: local tissucol application
  Arms: treatment with tissucol
Procedure: drainage system — application of vacuum drainage system
  Other Names: vacuum drainage system
  Arms: vacuum drainage system

SUMMARY:
The aim of this study is to demonstrate the efficacy of fibrin sealant (Tissucol-Baxter) in preventing pocket haematoma and subsequent complications in patients undergoing pacemaker or ICD implantation/replacement which cannot discontinue dual antiplatelet therapy (i.e. ASA and clopidogrel, ASA and prasugrel) or anticoagulant therapy (i.e. warfarin, heparin, low molecular weight heparin).

Fibrin-based sealant is available for local haemostasis. A recent study (Milic DJ et al, 2005 Europace, 7: 374-379) has shown the efficacy of the fibrin sealant in prevention of pacemaker pocket haematoma in 40 patients undergoing pacemaker implantation who are receiving anticoagulant treatment.

Patients with dual antiplatelet therapy (DAT) are prone to a high risk of bleeding during surgical procedures. Thus, the routine use is the discontinuation of DAT al least 4-7 days before the intervention. This practice may result in a high risk of thrombotic events in patients with coronary stenting.

Recently, in our Center we started the use of a fibrin sealant for local haemostasis (Tissucol Baxter), and the investigators observed a reduction in the incidence of pocket haematoma complication, the need of vacuum drainage system, and the reduction of hospital stay.

DETAILED DESCRIPTION:
Purpose of the study. The purpose of this study is to demonstrate the efficacy of a fibrin sealant (Tissucol-Baxter) in prevention pocket haematoma and subsequent complications in patients who required implantation/replacement of a pacemaker or ICD wich cannot discontinue dual antiplatelet or anticoagulant therapy.

Target. The primary endpoint is to test the impact of pocket haematoma in patients treated with tissucol compared to a conventional treatment with vacuum drainage system without dual antiplatelet or anticoagulant therapy discontinuation.

The secondary endpoint is to compare the length of hospitalization between the two groups.

Type of study. Prospective, randomized, single center, open label.

Materials and methods. Will be consecutively enrolled approximately 100 patients.

Inclusion criteria: patients over the age of eighteen who require an initial implantation or replacement of a device (pacemaker, biventricular pacemaker, ICD) treated with:

* dual antiplatelet therapy (clopidogrel or prasugrel or ticlopidine, and acetylsalicylic acid) or
* anticoagulants (warfarin or heparin or low molecular weight heparin). Patients Do not discontinue the antiplatelet or anticoagulant therapy.

According to a randomization list, patients will be assigned to tissucol treatment or vacuum drainage system:

* 50 patients: treated with local application of tissucol in the pocket of pacemaker/ICD;
* 50 patients: treated with vacuum drainage system.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require an initial implantation or replacement of a device (pacemaker, biventricular pacemaker, implantable cardiac defibrillator) treated with:

  * Dual antiplatelet therapy (i.e. ASA and clopidogrel, ASA and prasugrel) or
  * Anticoagulant therapy (warfarin, heparin, LMWH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Complications of pocket device: haematoma and bleeding.Pocket haematoma is defined as palpable swelling of the device pocket exceeding the size of the generator.Bleeding is defined as > 100 ml amount of fluid collected in the drainage system. | 45 days after intervention

SECONDARY OUTCOMES:
The duration of the hospital stay | 45 days after intervention
The number of outpatient visits following the hospitalization | 45 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Emilio V Dovellini, MD, Principal Investigator — Division of Invasive Cardiology, Careggi Hospital
Locations (1):
- Division of Invasive Cardiology 1, Careggi Hospital, Florence, Italy